CLINICAL TRIAL: NCT03623165
Title: An Observational, Prospective, Single Arm, Multi-Center Registry to Evaluate the Cordella™ Heart Failure System in New York Heart (NYHA) Class III Heart Failure Patients (PRODIGY Registry)
Brief Title: PRODIGY Registry in NYHA Class III Heart Failure Patients
Status: Terminated | Type: Observational
Why Stopped: same information will be collected in upcoming IDE trial
Sponsor: Endotronix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ETX-HFS-CHFS-01
Record Dates: First submitted 2018-06-27; First posted 2018-08-09 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure NYHA Class III
Keywords: Heart Failure; NYHA Class III
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm: Cordella™ Heart Failure System
  Interventions: Device: Cordella™ Heart Failure System

INTERVENTIONS:
Device: Cordella™ Heart Failure System — The Cordella™ Heart Failure System electronically transfers communications and data from a set of medical devices in a heart failure patient's home to a database for storage, retrieval, and display to healthcare providers.

SUMMARY:
This is an observational, prospective, single arm, multi-center registry to evaluate the Cordella™ Heart Failure System (CHFS) in up to 250 NYHA Class III HF patients .

DETAILED DESCRIPTION:
The subjects in this registry will participate in the Screening Visit, and Follow-Up Visits. After the Screening Visit, eligible subjects will be trained on at-home use of the CHFS to measure BP, HR, SpO2, weight and optional ECG.

They will be instructed to perform daily measurements of the parameters which will all be wirelessly transmitted to a secure website for review using the myCordella™ Patient Management Portal (PMP). Clinicians will be able to view Blood Pressure (BP), Heart Rate (HR), peripheral capillary oxygen saturation (SpO2), weight and Electrocardiogram (ECG) (optional) data through the myCordella™ PMP.

Subjects will return for follow up visits at 3, 6, and 12 months after enrollment or until study termination.

At Month 6, the primary endpoint will be assessed through evaluation of the subjects Quality of Life using the completed KCCQ Questions.

Assessment of secondary endpoints will be performed throughout the study duration, including evaluation of adverse events, and heart failure-related hospitalizations and medication changes. Additionally, Health Economics will be assessed per subject and per site via a detailed site questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent
2. Male or female complex CCM eligible patients or equivalent and at least 18 years of age
3. Diagnosis of HF ≥ 3 months and NYHA Class III HF at the time of Screening
4. Subject fluent in English (written and oral) and with sufficient eyesight, hearing, and mental capacity to respond to the Cordella™ Heart Failure System audio/visual cues and operate the Cordella™ Heart Failure System
5. Subject has sufficient Cellular and/ or Wi- Fi Internet coverage at home
6. Subject agrees:

   1. that the treating Investigator is their solely complex CCM physician
   2. to return to the treating Investigator for all scheduled follow up visits and can return to the hospital for follow up

Exclusion Criteria:

1. Subjects enrolled in another investigational trial.
2. Subjects who are unwilling or deemed by the Investigator to be unwilling to comply with the study protocol, or subjects with a history of non-compliance
3. Severe illness, other than heart disease, which would limit survival to <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in this study will be male or female Complex Chronic Care Management (CCM) eligible patients with a diagnosis of NYHA Class III heart failure. Subjects must be diagnosed with heart failure for a minimum of 3 months at time of screening.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) change from baseline to 6 month | Baseline- 6 month
  The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. For brevity, only the performance characteristics of the overall summary score are presented in this discussion.The answers patients give to the KCCQ's questions are used to calculate scores in ten scales: Physical Limitation, Symptom Stability, Symptom Frequency, Symptom Burden, Total Symptom, Social Limitation, Self-Efficacy, Quality of Life, Clinical Summary, Overall Summary

SECONDARY OUTCOMES:
Percentage of device success | 12 months post Enrollment
  Percentage of device success as documented by ability of the System to successfully transmit data (BP, HR, SpO2, weight and optional ECG) to a secure database.
Frequency of Adverse Events | 12 months post Enrollment
  Frequency and rates of adverse events(AEs) throughout the study
Heart Failure Hospitalizations | 12 months post Enrollment
  Number of HF hospitalizations, HF treatments in a hospital day-care setting, or urgent outpatient clinic HF visits
Device/system-related complications | 12 months post Enrollment
  Incidence of Device/system-related complications
Adherence to regular myCordella™ Peripherals measurements | 12 months post Enrollment
  Compliance in using myCordella™ at minimum 5 out of 7 days
Heart Failure Related Medication Changes | 12 months post Enrollment
  Changes to Heart Failure Related Medication from Baseline through 12 month post Enrollment
Health Economic Questionnaire & Cost Effectiveness Analysis | 12 months post Enrollment
  Cost Effectiveness of treating Complex Chronic Care Management (CCM) patients with Heart Failure using the Cordella™ Heart Failure System will be assessed with a questionnaire generated by a Health Economics expert from sponsor. Analyses will include: CCM billing practices, overall economic costs for: hospitalizations (including length of stay), treatment in day-care settings, treatment in urgent care, medication costs, as well as indriect costs (missed days at work, caregiver support, etc.)
Kansas City Cardiomyopathy Questionnaire (KCCQ) change from baseline to 12 month | 12 months post Enrollment
  The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. For brevity, only the performance characteristics of the overall summary score are presented in this discussion.The answers patients give to the KCCQ's questions are used to calculate scores in ten scales: Physical Limitation, Symptom Stability, Symptom Frequency, Symptom Burden, Total Symptom, Social Limitation, Self-Efficacy, Quality of Life, Clinical Summary, Overall Summary

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sauerland, Study Director — Endotronix, Inc.
Locations (4):
- United States (4):
  - USC Keck School of Medicine, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Craig Cardiovascular Center, Gonzales, Texas

IPD SHARING:
Plan to Share IPD: No